CLINICAL TRIAL: NCT01674868
Title: Pilot RCT of Fluoxetine vs Placebo to Treat Motor, Language and Unilateral Neglect After Ischemic Stroke
Brief Title: Fluoxetine for Motor, Aphasia, and Neglect Recovery After Ischemic Stroke
Acronym: FLAN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to find patients meeting inclusion/exclusion criteria
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Randie Black-Schaffer MD, Medical Director, Stroke Program, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLAN SpauldingRH
Record Dates: First submitted 2012-08-24; First posted 2012-08-29 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Stroke
Keywords: stroke; recovery; fluoxetine; aphasia; neglect; motor
MeSH Terms: conditions — Stroke; Aphasia | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluoxetine (Experimental): Subjects will take 20 mg fluoxetine daily for 90 days after stroke
  Interventions: Drug: fluoxetine
- placebo (Placebo Comparator): Subjects will take one pill daily for 90 days after stroke.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fluoxetine — 20 mg daily for 90 days starting day 5-10 after stroke.
  Arms: Fluoxetine
Drug: placebo — subjects will take one pill po daily for 90 days.
  Arms: placebo

SUMMARY:
This pilot study will recruit 25 subjects to assess the feasibility of replicating the FLAME study (Chollet, et al. Lancet 2011), a randomized controlled trial (RCT) that assessed the effect of fluoxetine vs placebo on motor recovery after ischemic stroke, in an American sample of post-acute stroke patients. This trial will in addition examine the effect of treatment with fluoxetine versus placebo on concurrent deficits in language and hemispatial attention, as well as post-stroke fatigue and will evaluate the durability of observed effects. The results of this pilot trial will be used to develop power estimates for a larger trial and to evaluate recruitment and intervention completion rates for subjects in an American post-acute environment. There are two additional substudies: the first will use MRI to assess structural changes at the beginning and end of the intervention; the second will examine the relationship of serum biomarkers of inflammation to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic infarction within 15 days
* Admission NIHSS item 5 score equal to or >2 -Able to give informed consent, with surrogate consent acceptable-

Exclusion Criteria:

* Pre-stroke modified Rankin Scale score equal or .3
* Pregnant or lactating
* Taking an SSRI on admission to SRH
* Taking a medication likely to have adverse interaction with an SSRI
* Unable to return for follow-up testing days 90,180
* Concurrent medial condition likely to worsen patient's functional status over next 6 months
* Unable to competently participate in testing for 45min-2hrs with rest breaks
* for MRI substudy: contraindication to MRI

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Motor Scale (FMMS) | baseline to 90 days
  change in FMMS score
Fugl-Meyer Motor Scale (FMMS) | baseline to 180 days
  change in FMMS

SECONDARY OUTCOMES:
Western Aphasia Battery | baseline to 90 days
  change in Western Aphasia Quotient
Behavioral Inattention Test (BIT) | baseline to 90 days
  change in BIT
Behavioral Inattention Test (BIT) | baseline to 180 days
  change in BIT
Functional Independence Measure | baseline to discharge
  change in FIM
Fatigue Severity Scale | baseline to 90 days
Beck Depression Inventory | baseline to 90 days
Western Aphasia Battery | baseline to 180 days
  change in Western Aphasia Quotient
Beck Depression Inventory | baseline to 180 days
Fatigue Severity Scale | baseline to 180 days
modified Rankin Scale | baseline to 90 days
modified Rankin Scale | baseline to 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States